CLINICAL TRIAL: NCT00003623
Title: Megadose Vitamins as Chemoprevention of Transitional Cell Carcinoma of the Bladder
Brief Title: High-Dose Multivitamins Compared to a Placebo in Preventing the Recurrence of Cancer in Patients With Early Stage Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCCTG-979252; CDR0000066702 (Registry Identifier: PDQ (Physician Data Query)); NCI-P98-0138
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Bladder Cancer
Keywords: recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multivitamin (Experimental): Patients receive multivitamins orally once daily for 3 years. Patients are followed every 3 months for 2 years, then every 6 months for 1 year, and then annually thereafter.
  Interventions: Dietary Supplement: multivitamin
- Placebo (Placebo Comparator): Patients receive placebo orally once daily for 3 years. Patients are followed every 3 months for 2 years, then every 6 months for 1 year, and then annually thereafter.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: multivitamin
  Arms: Multivitamin
Other: Placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of high-dose multivitamins may be an effective way to prevent the recurrence of early stage bladder cancer. It is not yet known whether high-dose vitamins are more effective than no further therapy in decreasing the risk of early-stage bladder cancer.

PURPOSE: Randomized double-blinded phase III trial to compare the effectiveness of high-dose multivitamins with a placebo in preventing the recurrence of cancer in patients with early stage bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVE: I. Determine whether high dose multivitamins have chemopreventive efficacy beyond standard therapy in reducing the risk of recurrence in patients with resected stage 0 and I (Ta, T1, and Tis) transitional cell carcinoma of the bladder.

OUTLINE: This is a randomized, double blind study. Patients are randomized to receive multivitamins or placebo orally once daily for 3 years. Patients are followed every 3 months for 2 years, then every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage 0 and I (Ta, T1 or Tis) resected transitional cell carcinoma of the bladder No advanced disease or muscle invasion No history of transitional cell carcinoma of the prostate

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Greater than 3 years Hematopoietic: WBC at least 3500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 3 times ULN SGOT no greater than 3 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: Not pregnant or nursing Fertile patients must use effective contraception At least 5 years since prior malignancy except nonmetastatic squamous cell or basal cell carcinoma of the skin No history of drug interactions which could affect therapy No immunodeficiency

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior intravesical BCG required (if T1 or Tis pathology and negative cytology PAB) Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the pelvis Surgery: Not specified Other: Intravesical therapy within 30 days allowed At least 30 days since greater than 2 multivitamins daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1999-10; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Prevention of reoccurence of early stage bladder cancer | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Blute, MD, Study Chair — Mayo Clinic
Locations (17):
- United States (16):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada